CLINICAL TRIAL: NCT05017285
Title: A Multicentre Randomised Controlled Trial Evaluating the Benefit of Median Lobe Preservation on the Incidence of Retrograde Ejaculation During Prostate Enucleation by HoLEP.
Brief Title: Ejaculation Preservation After Laser Enucleation Prostate
Acronym: EPALEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-A00031-40
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: A prospective randomised multicentre single-blind comparative study of two parallel groups of patients scheduled for HoLEP prostate resection:
  Group 1 Conventional HoLEP prostate resection procedure with enucleation of all three lobes (3-lobe, 2-lobe or monobloc technique).
  Group 2 Enucleation of the lateral lobes and preservation of the medial tissue between the bladder neck and Veru montanum Each patient will be evaluated five times during the study (D0, M1, M3, M6, M12) The total duration of the study is 2 years (1 year of recruitment and 1 year of follow-up).
Who Masked: Participant
Masking Description: The patient does not know which type of surgery is used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HoLEP classic (Other): Standard HoLEP prostate resection procedure with enucleation of all three lobes (3-lobe, 2-lobe or monobloc technique).
  Interventions: Procedure: HoLEP classic
- HoLEP with median lobe preservation (Experimental): Enucleation of the lateral lobes and preservation of the medial tissue between the bladder neck and Veru montanum.
  Interventions: Procedure: HoLEP with median lobe preservation

INTERVENTIONS:
Procedure: HoLEP with median lobe preservation — Enucleation of the lateral lobes and preservation of the medial tissue between the bladder neck and Veru montanum
  Arms: HoLEP with median lobe preservation
Procedure: HoLEP classic — Standard HoLEP prostate resection procedure with enucleation of all three lobes (3-lobe, 2-lobe or monobloc technique).
  Arms: HoLEP classic

SUMMARY:
A multicentre randomised controlled trial evaluating the benefit of median lobe preservation on the incidence of retrograde ejaculation during prostate enucleation by HoLEP.

DETAILED DESCRIPTION:
The main objective of the study is to compare the incidence of retrograde ejaculation at 6 months in patients undergoing Holep surgery for prostatic adenoma according to two randomized surgical techniques: conventional surgical procedure of removal of the 3 prostatic lobes versus preservation of the median lobe.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years and older who have signed their consent to participate in the study
* Patient with preserved cognitive functions
* Patient with BPH characterised by an IPSS score ≥ 12, a Qmax ≤ 15 ml/s and an ultrasound-assessed prostate volume between 40 and 150 cc
* Patient for whom an indication for prostatic resection by HoLEP has been made,
* A patient who is sexually active and willing to maintain sexual activity after surgery
* Patient affiliated to a social security system or beneficiary of such a system

Exclusion Criteria:

* History of prostate surgery or prostate radiotherapy
* Urethral stenosis
* Cancer or a history of cancer
* Patient with a life expectancy of less than 2 years
* Patient refusing partial surgery
* History of vasectomy, erectile dysfunction or ejaculation
* Mental deficiency or any other reason that may hinder the understanding or the strict application of the protocol
* Patient under court protection, guardianship or curatorship
* Patient already included in another therapeutic study protocol or having participated in another trial in the previous three months

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study on prostate hyperplasia
Enrollment: 11 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Retrograde ejaculation | Month 6
  Existence of retrograde ejaculation at Month 6, as evidenced by the presence of spermatozoa in the urine following sexual intercourse (as evidenced by an ECBU performed within 24 hours of intercourse)

SECONDARY OUTCOMES:
International Prostate Symtom Score (IPSS) assessment | Month 1
  The International Prostate Symtom Score (IPSS) is a structured and validated self-administered questionnaire that assesses the intensity and discomfort of lower urinary tract disorders. It consists of 7 questions on symptomatology with answers rated from 0 to 5 and one question on quality of life. A score of <7 is mild, a score of 8-19 is moderate and a score of >20 is severe
International Prostate Symtom Score (IPSS) assessment | Month 3
  The International Prostate Symtom Score (IPSS) is a structured and validated self-administered questionnaire that assesses the intensity and discomfort of lower urinary tract disorders. It consists of 7 questions on symptomatology with answers rated from 0 to 5 and one question on quality of life. A score of <7 is mild, a score of 8-19 is moderate and a score of >20 is severe
International Prostate Symtom Score (IPSS) assessment | Month 6
  The International Prostate Symtom Score (IPSS) is a structured and validated self-administered questionnaire that assesses the intensity and discomfort of lower urinary tract disorders. It consists of 7 questions on symptomatology with answers rated from 0 to 5 and one question on quality of life. A score of <7 is mild, a score of 8-19 is moderate and a score of >20 is severe
International Prostate Symtom Score (IPSS) assessment | Month 12
  The International Prostate Symtom Score (IPSS) is a structured and validated self-administered questionnaire that assesses the intensity and discomfort of lower urinary tract disorders. It consists of 7 questions on symptomatology with answers rated from 0 to 5 and one question on quality of life. A score of <7 is mild, a score of 8-19 is moderate and a score of >20 is severe
Men Sexual Health Questionnaire (MSHQ) score assessment | Month 3
  The Men Sexual Health Questionnaire (MSHQ) assesses a patient's ability to have sex. It consists of 25 questions that explore the ability to have erections, the quality of ejaculations and the satisfaction felt during intercourse and sexual desire.
  The total score (16 to 125 points maximum) is broken down into 6 sub-scores that explore erection (0 to 15 points), discomfort with erection problems (1 to 5 points), ejaculation (1 to 35 points), discomfort with ejaculation problems (1 to 5 points), satisfaction (6 to 30 points), sexual activity and desire (7 to 35 points)
Men Sexual Health Questionnaire (MSHQ) score assessment | Month 6
  The Men Sexual Health Questionnaire (MSHQ) assesses a patient's ability to have sex. It consists of 25 questions that explore the ability to have erections, the quality of ejaculations and the satisfaction felt during intercourse and sexual desire.
  The total score (16 to 125 points maximum) is broken down into 6 sub-scores that explore erection (0 to 15 points), discomfort with erection problems (1 to 5 points), ejaculation (1 to 35 points), discomfort with ejaculation problems (1 to 5 points), satisfaction (6 to 30 points), sexual activity and desire (7 to 35 points)
Men Sexual Health Questionnaire (MSHQ) score assessment | Month 12
  The Men Sexual Health Questionnaire (MSHQ) assesses a patient's ability to have sex. It consists of 25 questions that explore the ability to have erections, the quality of ejaculations and the satisfaction felt during intercourse and sexual desire.
  The total score (16 to 125 points maximum) is broken down into 6 sub-scores that explore erection (0 to 15 points), discomfort with erection problems (1 to 5 points), ejaculation (1 to 35 points), discomfort with ejaculation problems (1 to 5 points), satisfaction (6 to 30 points), sexual activity and desire (7 to 35 points)
International Index of Erectil Function (IIEF-5) score assessment | Month 3
  The IIEF-5 (International Index of Erectile Function) questionnaire consists of 5 questions that assess erectile function over the past 6 months. Severe erectile dysfunction corresponds to a score of 5-10, moderate erectile dysfunction to a score of 11-15 and mild erectile dysfunction to a score of 16-20. A score of 21 to 25 corresponds to normal erectile function and scores between 1 and 4 are not interpretable.
International Index of Erectil Function (IIEF-5) score assessment | Month 6
  The IIEF-5 (International Index of Erectile Function) questionnaire consists of 5 questions that assess erectile function over the past 6 months. Severe erectile dysfunction corresponds to a score of 5-10, moderate erectile dysfunction to a score of 11-15 and mild erectile dysfunction to a score of 16-20. A score of 21 to 25 corresponds to normal erectile function and scores between 1 and 4 are not interpretable.
International Index of Erectil Function (IIEF-5) score assessment | Month 12
  The IIEF-5 (International Index of Erectile Function) questionnaire consists of 5 questions that assess erectile function over the past 6 months. Severe erectile dysfunction corresponds to a score of 5-10, moderate erectile dysfunction to a score of 11-15 and mild erectile dysfunction to a score of 16-20. A score of 21 to 25 corresponds to normal erectile function and scores between 1 and 4 are not interpretable.
Urine flow (Qmax) measurement | Month 1
  Assessment of urine flow (Qmax) by ultrasound
Urine flow (Qmax) measurement | Month 3
  Assessment of urine flow (Qmax) by ultrasound
Urine flow (Qmax) measurement | Month 6
  Assessment of urine flow (Qmax) by ultrasound
Urine flow (Qmax) measurement | Month 12
  Assessment of urine flow (Qmax) by ultrasound
Adverse events related to the procedure | Month 12
  Presence of urinary incontinence and occurrence of adverse events related to the procedure
Assessment of resected volume / total volume | Month 12
  Assessment of resected volume / total volume assessed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BALDINI, MD PD, Principal Investigator — Clinique de la Sauvegarde
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No